CLINICAL TRIAL: NCT06482840
Title: Safety and Efficacy of EasyCool Catheter - Prospective Monocentric Study
Brief Title: Safety and Efficacy of EasyCool Catheter
Status: Active, not recruiting | Type: Observational
Sponsor: MedFact Engineering GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: CT04-01_EasyCool
Record Dates: First submitted 2024-06-26; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Cardiac Arrhythmia
Keywords: EasyCool Catheter; cardiac ablation
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about risks and benefit of EasyCool Catheter for cardiovascular ablation in real-world patients suffering from cardiac arrythmias.

The main question[s] it aims to answer are:

* will the cardiac arrythmia be removed and remain absent oc recurrent also 3 months after procedure
* what are the adverse events at procedure, after 3 and 6 months

All participants will receive cardiac ablation with EasyCool catheter.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring intracardial RF- Ablation with irrigated catheter

Exclusion Criteria:

* Absence of patient´s consent;
* Age <12 years;
* Pregnancy or breast-feeding women;
* Acute local infection;
* Acute systemic infection;
* Atrial thrombosis or myxoma - the transseptal approach is contraindicated in patients with left atrial thrombus;
* Existence of active Implants (Pacemaker, Defibrillator etc.);
* Hemodynamic instability;
* Hypercoagulability;
* Inadequate tissue damaged e.g. by radiation or suppuration;
* Obstruction of the artery or vein selected for insertion;
* Patients with artificial heart valve: the use of intracardial catheters is not advised;
* Physiologic or anatomic abnormalities that could cause postoperative complications e.g. aneurysms in the application area, bleeding diathesis, decreased resistance to infections;
* Previously diagnosed spasms of the coronary arteries;
* Recurrent metastasizing cancer;
* Sepsis;
* Severe concomitant illness for which an increase or surgery time is associated with a significant increased risk;
* Thrombosis of the leg veins and the deep pelvic vein.

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Intracardial RF-Ablation procedure at following indications:
  * Atrial Tachycardia
    * Tricuspid istmus flutter
    * Atypical flutter
    * Focal atrial tachycardia
    * Atrial fibrillation
  * AV-node re-entrant tachycardia;
  * Tachycardia heart rhythm disturbances associated with accessory pathways;
  * Ventricular Tachycardia.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2023-12-08 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Removal of treated cardiac arrythmia | 3 months after procedure
  Removal of treated cardiac arrhythmia and absence of recurrence of the arrythmia

SECONDARY OUTCOMES:
Adverse Events | at procedure, after 3 and 6 months
  all adverse events in context to procedure and product

CONTACTS AND LOCATIONS:
Overall Officials: Abdeddayem Haggui, Prof, Principal Investigator — Centre Hospitalier International de Carthagène, Tunisia
Locations (1):
- Centre Hospitalier International de Carthagène, Tunis, Centre Urbain Nord, Tunisia